CLINICAL TRIAL: NCT02444416
Title: Prospective Registry of Acute Heart Failure
Status: Recruiting | Type: Observational
Sponsor: Sebastian Carballo (Other)
Responsible Party: Sponsor-Investigator, Sebastian Carballo, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: 14-019
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Acute Heart Failure
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: blood sample

SUMMARY:
Context:

Heart failure is associated with a high morbidity and mortality rate and represents a significant worldwide public health burden. In European countries, the total amount of the expenses related to heart failure represents 1 to 2% of the total health budget with 75% spent during hospitalizations, making heart failure the most expensive pathology in cardiology. Acute heart failure (AHF) has a poor prognosis despite improvements in therapy. Hospital mortality is 2 to 4% the risk of death or readmission in the six months following hospitalization is high.

Patients hospitalized for heart failure represent a very heterogeneous population in terms of etiologies, clinical presentations and/or co-morbidities. Consequently, this implies variable outcomes in terms of morbidity and mortality, probably due to their different prognostic factors. The precise spectrum of etiologies and prognostic factors of AHF in non selected populations has not been exhaustively studied and only a few predictive models concerning AHF have been validated.

Ischemic heart disease, valvulopathy, arrhythmias, infections, hypertension and lack of therapeutic compliance are often quoted as being the factors triggering heart failure. Some triggering factors (ischemic heart disease, pulmonary infections, acute renal failure) seem to be strongly associated with a poor prognosis in terms of hospital/out-patient mortality and re-hospitalization rate.

The complex relation between heart failure and acute renal failure is defined by the cardio-renal syndrome. Thirty percent of patients hospitalized for AHF will be diagnosed with an acute renal failure at admission or with worsening kidney failure during hospitalization. It seems that heart failure and cardio-renal syndrome are two distinct entities with a different prognosis. The type of acute renal failure (functional, renal or post-renal) in these patients and the prognostic value of these etiologies is still not firmly established.

A thorough determination of the etiologies and prognostic factors of AHF are necessary in order to allow the identification of high-risk patients and the improvement of heart failure management.

Objectives:

* To create an observational registry of all patients hospitalized for a AHF
* To determine the precise prevalence of etiologies and the prognostic factors of AHF in a non selected population. Among the prognostic factors, to establish the specific role of acute renal failure
* To establish the optimal initial assessment of patients hospitalized for heart failure
* To validate and compare with prospective data the results of a retrospective cohort study carried out at the University Hospital of Geneva who established the re-hospitalization and mortality outcome of patients hospitalized for heart failure.

Method:

Creation of an observational registry associated with a biobank including patients hospitalized for AHF in the Department of General Internal medicine (SMIG) and in the Departments of Specialties at the University Hospital of Geneva.

Anticipated results:

* To identify the prevalence of the etiologies and the prognostic factors of the heart failure
* To establish the optimal initial assessment of the patients hospitalized for a heart failure. Among the prognostic factors, to establish the specific role of acute renal failure
* To validate and compare results of a retrospective cohort study carried out at the University Hospital of Geneva which established the re-hospitalization and mortality outcome of patients hospitalized AHF
* To improve the management of hospitalized patients with AHF with a robust identification of the etiologies and a better identification of high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Usual clinical presentation of acute heart failure as defined by the European Society of Cardiology : Gradual onset or new or worsening symptoms of rapid heart failure (eg, dyspnea, edema of the lower limbs and tiredness ) and signs of heart failure (eg elevation of jugular venous pressure, crackles, moving the shock peak) requiring urgent treatment.
* Brain natriuretic peptide or value of brain natriuretic peptide (BNP) greater than 100 ng / L.

Exclusion Criteria:

* Inability or refusal to consent to participate in the study cohort.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized for an acute heart failure
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2014-12; Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence of different clinical presentations of the acute heart failure | baseline
Prevalence of the triggers of the acute heart failure | baseline
Prognostic factors (including the acute renal failure and worsening renal function) in the acute heart failure | baseline
Rehospitalization and early and late mortality | 30 days, 90days, 1 year and 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Derived] Carballo D, Garin N, Stirnemann J, Mamin A, Prendki V, Meyer P, Marti C, Mach F, Reny JL, Serratrice J, Kaiser L, Carballo S. Prognosis of Laboratory-Confirmed Influenza and Respiratory Syncytial Virus in Acute Heart Failure. J Clin Med. 2021 Sep 30;10(19):4546. doi: 10.3390/jcm10194546. PMID 34640562
- [Derived] Carballo D, Stirnemann J, Garin N, Marti C, Serratrice J, Carballo S. Eligibility for sacubitril-valsartan in patients with acute decompensated heart failure. ESC Heart Fail. 2020 Jun;7(3):1282-1290. doi: 10.1002/ehf2.12676. Epub 2020 Mar 13. PMID 32167679
- [Derived] Carballo S, Musso P, Garin N, Muller H, Serratrice J, Mach F, Carballo D, Stirnemann J. Prognostic Value of the Echocardiographic Probability of Pulmonary Hypertension in Patients with Acute Decompensated Heart Failure. J Clin Med. 2019 Oct 15;8(10):1684. doi: 10.3390/jcm8101684. PMID 31618841